CLINICAL TRIAL: NCT05642390
Title: Prospective Observational Study About SEBBIN Silicone Gel-filled INTEGRITY Mammary Implants
Brief Title: SEBBIN INTEGRITY Round Implants
Status: Terminated | Type: Observational
Why Stopped: sponsor's strategic decision
Sponsor: Groupe SEBBIN (Industry)
Responsible Party: Sponsor
Other Study IDs: PEC 20-08-001
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Complication; Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure | interventions — Breast Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Breast implant — Patients operated for breast augmentation or reconstruction.

SUMMARY:
This study is part of the clinical evaluation of SEBBIN silicone gel-filled INTEGRITY implants, included in the technical file of the device. The aim of the study is to gather additional data about the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18-year-old.
* The patient is a woman.
* The patient was prescribed with a surgery for a breast augmentation or reconstruction, unilaterally or bilaterally with silicone gel-filled SEBBIN INTEGRITY mammary implants.
* The patient has been informed of the study, has read the patient information letter and provided consent in writing.

Exclusion Criteria:

* The patient is pregnant or breastfeeding.
* The patient has silicone implants somewhere else than in the breast.
* The patient was diagnosed with one of the following pathologies:

  * Systemic lupus erythematous, Sjogren syndrome, scleroderma, polymyositis, or any other connective tissue disease.
  * Rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, or any other inflammatory arthritic disease.
  * Arthritis, fibromyalgia, chronic fatigue syndrome, or any other mechanic or degenerative non-inflammatory rheumatic disease.
  * History of implant-associated anaplastic large cell lymphoma (BIA-ALCL).
  * Symptomatic autoimmune disease.
* The patient has a pathology that could delay healing (does not apply to the reconstruction group).
* The patient has cancer (does not apply to the reconstruction group).
* The patient has anatomical or physiological conditions that could lead to postoperative complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Study Population: The study population will be recruited from prospective adult patients operated for breast augmentation or reconstruction, unilaterally or bilaterally with SEBBIN silicone gel filled INTEGRITY mammary implants.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Complication rate | At 10 years of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- SEBBIN, Saint-Ouen-l'Aumône, France